CLINICAL TRIAL: NCT07085299
Title: Correlation Study Between Gut Microbiota and Prognosis in Patients With Intracranial Arterial Stenosis（GROW-ICAS）
Brief Title: Gut Microbiota and Prognostic Outcomes in Intracranial Arterial Stenosis Patients（GROW-ICAS）
Status: Recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: GROW-ICAS
Record Dates: First submitted 2025-07-01; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-06

CONDITIONS: Intracranial Artery Stenosis
Keywords: intracranial artery stenosis; Gut Microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
GROW-ICAS (Gut microBiota and prOgnostic Outcomes in IntraCranial Arterial Stenosis) is a prospective observational cohort study that enrolls patients with intracranial arterial stenosis to investigate the correlations between their gut microbiota, metabolomic, and transcriptomic profiles and three key clinical domains: functional outcomes, vascular plaque imaging characteristics, and post-stroke non-motor dysfunctions (including cognitive impairment, depression, anxiety, and fatigue).

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-80 years.
2. Intracranial arterial stenosis confirmed by CTA/MRA/DSA.
3. Local residency ≥6 consecutive months.
4. Signed informed consent.

Exclusion Criteria:

1. Tandem extracranial stenosis (≥50%) proximal to the target intracranial stenotic vessel.
2. Non-atherosclerotic intracranial stenosis.
3. Extracranial/intracranial endovascular treatment within 30 days pre-enrollment or planned intervention within 6 months.
4. Intracranial hemorrhage within 90 days pre-enrollment.
5. Pre-existing intracranial tumor, cerebral aneurysm, or arteriovenous malformation.
6. Cardioembolic embolism.
7. Active bleeding/hemorrhagic diathesis.
8. Major surgery within 30 days pre-enrollment or planned within 6 months post-enrollment.
9. Severe neurological deficits impairing independent living or dementia/psychiatric disorders hindering follow-up.
10. Pregnancy/lactation/planned pregnancy.
11. Chronic inflammatory/autoimmune diseases.
12. Uncontrolled hypertension or diabetes.
13. Severe cardiac/hepatic/renal dysfunction, hematologic disorders, malignancy, or life expectancy <1 year.
14. MRI contraindications.
15. History of depression/anxiety/cognitive impairment requiring therapy.
16. Antibiotic/probiotic/glucocorticoid/immunosuppressant use within 1 month pre-enrollment.
17. Current/planned participation in other trials.
18. Inability to cooperate due to psychiatric/emotional disorders.
19. Other investigator-deemed ineligibility.

Ages: 30 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with intracranial arterial stenosis recruited from the Department of Neurology, Nanjing First Hospital (Affiliated Nanjing Hospital of Nanjing Medical University)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Stroke Recurrence in Patients with Symptomatic Intracranial Arterial Stenosis | From enrollment to 1 year
  Patients with symptomatic intracranial arterial stenosis experiencing recurrent cerebrovascular events, defined as either novel ischemic stroke or transient ischemic attack (TIA).
Stroke Occurrence in Patients with Asymptomatic Intracranial Arterial Stenosis | From enrollment to 1 year
  Incident cerebrovascular events-comprising ischemic stroke or transient ischemic attack (TIA)-occurring in patients exhibiting asymptomatic intracranial arterial stenosis.

SECONDARY OUTCOMES:
Changes in Imaging Characteristics of Intracranial Vascular Plaques. | From enrollment to 1 year
  * Plaque Burden = Σ (Cross-sectional wall area - Cross-sectional lumen area) / Σ Cross-sectional wall area × 100%
  * Change in Plaque Burden = Plaque burden at Week 24/48 - Baseline plaque burden

OTHER OUTCOMES:
Functional outcomes were assessed using the modified Rankin Scale (mRS). | From enrollment to 1 year
  Functional outcomes were assessed using the modified Rankin Scale (mRS), a 7-point scale ranging from 0 to 6, with higher scores indicating greater disability.
Cognitive function was assessed using the Mini-Mental State Examination (MMSE) and Montreal Cognitive Assessment (MoCA). | From enrollment to 1 year
  Both scales have a maximum score of 30 points, with lower scores indicating greater cognitive impairment.
Fatigue severity was assessed using the 9-item Fatigue Severity Scale (FSS). | From enrollment to 1 year
  The FSS is a valid and reliable 7-point Likert scale used for assessing and quantifying fatigue, with scores ranging from 1 (strongly disagree) to 7 (strongly agree). A higher score indicates more severe fatigue.
Depression severity was assessed using the 17-item Hamilton Depression Rating Scale (HAMD). | From enrollment to 1 year
  The HAMD total score serves as a reliable indicator of symptom severity, where lower scores correspond to milder symptoms and higher scores indicate greater symptom severity.
Anxiety severity was assessed using the 14-item Hamilton Anxiety Rating Scale (HAMA). | From enrollment to 1 year
  The Hamilton Anxiety Rating Scale (HAMA-14) was administered to quantify anxiety severity. A direct correlation exists between total scores and clinical symptom burden, with elevated scores denoting increased severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No